CLINICAL TRIAL: NCT01280708
Title: Establishment of a National Thematic Network in Urology for the Extension of the Cohort DIVAT (Données Informatisées et Validées en Transplantation) in Surgical Parameters of Renal and Pancreatic Transplant Patients : An Innovative Tool for the Promotion of Epidemiological Studies, Identification of Risk Factors and Good Practices in the Domain of Transplant Surgery
Brief Title: Protocol DIVAT-Uro
Status: Terminated | Type: Observational
Why Stopped: This database did not have the desired inclusions or results and is therefore not sufficiently usable. This base is therefore abandoned in favor of a base on the pancreas much more promising both nationally and internationally.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/09/11-E
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2011-09

CONDITIONS: Kidney Transplantation; Pancreas-kidney Transplantation
Keywords: Urology; Nephrology; Renal and pancreas transplantation; Data base; Epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Capture data
  Interventions: Other: Capture data

INTERVENTIONS:
Other: Capture data — Capture and standardization of data of patients aged over 18 years received a kidney transplant or a simultaneous pancreas-kidney transplant from data sources will be performed by clinical research associates.The quality of data will be validated by cross annual audits. The statistical analysis will be made on a case by case according to clinical objectives.

SUMMARY:
The aim of project DIVAT-URO (Données Informatisées et Validées en Transplantation - Urology) is to organize a thematic network in urology traced on NetWork DIVAT to supplement the medical and biological data of DIVAT existing cohort with parameters of surgical transplantation of kidney and pancreas. These data will concern the transplantation itself and the events and complications related to surgery occurring throughout the follow-up. The collection will involve patients in the cohort DIVAT and future patients. This project will allow us to have the sufficiency of surgical transplantation by increasing the quantity and quality of information gathered thus avoiding the biases commonly upbraided against the retrospective studies. Finally, by supplementing it with new parameters, it will strengthen the medical and scientific interest of the cohort DIVAT and will open new perspectives for clinical trials in surgery and work in epidemiology.Networking of urologists and the expansion of the base DIVAT would carry out research in epidemiology and factors that may play a role in the outcome of renal and pancreatic transplantation. It would also help to define good practices. The first study from the proposed network DIVAT-Uro is assessing the impact of vesico-ureteric reflux on the occurrence of urinary tract infections and effects on survival of the transplant in the recipient adult.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Patients received a kidney transplant or a simultaneous pancreas-kidney transplant
* Patients who read the newsletter and signed the consent form on the computerization of data

Exclusion Criteria:

* Patients aged under 18 years
* Patients who did not sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years received a kidney transplant or a simultaneous pancreas-kidney transplant.
Sampling Method: Non-Probability Sample
Enrollment: 1616 (Actual)
Dates: Start 2012-01-02 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georges KARAM, Profesor, Principal Investigator — Nantes University Hospital; Lionel BADET, Profesor, Study Chair — Hospices Civils de Lyon; François IBORRA, Doctor, Study Chair — CHU de Montpellier; Jacques HUBERT, Profesor, Study Chair — Central Hospital, Nancy, France; Arnaud MEJEAN, Profesor, Study Chair — Hôpital Necker - AP-HP; Pascal RISCHMANN, Profesor, Study Chair — University Hospital, Toulouse
Locations (1):
- Nantes University Hospital, Nantes, France